CLINICAL TRIAL: NCT07326137
Title: A Prospective Observational Study of First-Line Systemic Therapy Combined With Celiac Plexus Blockade in Patients With Advanced Biliopancreatic Malignancies and Cancer-Related Pain
Brief Title: A Prospective Observational Study of First-Line Systemic Therapy Combined With Celiac Plexus Blockade for Advanced Biliopancreatic Cancer With Pain
Status: Recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Wan-Guang Zhang, Professor, Tongji Hospital
Other Study IDs: TJ-IRB202512171
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-12

CONDITIONS: Advanced Biliary Tract Cancer(BTC); Advanced Pancreatic Cancers; Cancer-related Pain
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Advanced Biliary Tract Cancer Cohort: Patients with histologically confirmed advanced biliary tract cancer (including cholangiocarcinoma) who are scheduled to receive first-line systemic therapy combined with celiac plexus neurolysis (CPN) for cancer-related pain.
  Interventions: Drug: First-Line Systemic Therapy; Procedure: Celiac Plexus Neurolysis (CPN)
- Advanced Pancreatic Cancer Cohort: Patients with histologically confirmed advanced pancreatic cancer (including pancreatic ductal adenocarcinoma) who are scheduled to receive first-line systemic therapy combined with celiac plexus neurolysis (CPN) for cancer-related pain.
  Interventions: Drug: First-Line Systemic Therapy; Procedure: Celiac Plexus Neurolysis (CPN)

INTERVENTIONS:
Drug: First-Line Systemic Therapy — Standard first-line systemic therapy regimens for advanced biliopancreatic malignancies, administered according to clinical guidelines. For biliary tract cancer, this may include regimens such as Durvalumab or Pembrolizumab combined with Gemcitabine and Cisplatin. For pancreatic cancer, this may include FOLFIRINOX or mFOLFIRINOX regimens, or Gemcitabine-based combinations. The specific regimen is determined by the treating physician based on the patient's cancer type, performance status, and standard of care.
Procedure: Celiac Plexus Neurolysis (CPN) — An interventional pain management procedure performed under CT or ultrasound guidance. It involves the injection of a neurolytic agent (such as absolute ethanol or 10% phenol) into the celiac plexus to block the transmission of pain signals from the upper abdomen. This procedure is intended to provide long-term pain relief for patients with advanced biliopancreatic malignancies.

SUMMARY:
This study is for patients with advanced bile duct or pancreatic cancer who are experiencing pain from their disease. The purpose of this research is to learn about the effects of combining a standard pain relief treatment (Celiac Plexus Block) with standard first-line cancer drugs.

Patients in this study will receive the Celiac Plexus Block procedure, which is intended to reduce pain, and will then begin their standard cancer medication regimen. Researchers will observe and compare how well this combined approach works to control pain and the cancer itself, and will monitor for any side effects. Participation in this study involves being followed by the research team for up to 2 years to track health outcomes.

The goal is to see if starting cancer treatment together with this specialized pain management technique is more helpful for patients compared to what is already known about the standard treatments alone.

DETAILED DESCRIPTION:
This is a prospective, observational, single-center cohort study designed to evaluate the clinical outcomes of integrating celiac plexus neurolysis (CPN) with standard first-line systemic therapy in patients diagnosed with advanced biliopancreatic malignancies and concomitant cancer-related pain.

Eligible participants are adults with histologically confirmed, inoperable advanced biliary tract cancer or pancreatic cancer, who present with moderate to severe abdominal pain and are candidates for first-line systemic treatment. All patients will be managed according to routine clinical practice; the decision to perform CPN and the choice of specific systemic therapy regimen will be determined by the treating physician team based on standard guidelines and individual patient circumstances, not by the study protocol.

The primary objective is to assess the efficacy of this integrated approach, with co-primary endpoints of pain response rate and objective tumor response rate. Pain response is defined as a reduction of ≥2 points in the Numeric Rating Scale score or a ≥50% decrease in opioid consumption sustained for ≥4 weeks. Tumor response will be evaluated per RECIST 1.1 criteria. Secondary objectives include comparing overall survival, progression-free survival, and quality of life metrics between the cohort receiving CPN combined with systemic therapy and a contemporary control cohort receiving systemic therapy alone. Safety will be assessed by monitoring the incidence and severity of adverse events related to both CPN and the systemic treatments.

Clinical data, including pain scores, analgesic usage, tumor imaging assessments, and laboratory results, will be prospectively collected at predefined time points for a follow-up period of up to 2 years. The study aims to provide real-world evidence on whether the early integration of interventional pain management with oncological treatment can improve overall patient outcomes in this population with high symptom burden.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced biliopancreatic malignancy (including biliary tract cancer or pancreatic cancer).
* Cancer-related pain: Baseline Numeric Rating Scale (NRS) pain score ≥ 4 points for over 1 week, with plans to receive celiac plexus neurolysis (CPN).
* Scheduled to receive a first-line systemic treatment regimen (e.g., PD-1/PD-L1 inhibitor monotherapy or in combination with chemotherapy/targeted therapy).
* ECOG Performance Status of 0-2 and an estimated life expectancy of ≥ 3 months.

Exclusion Criteria:

* Previous history of celiac plexus neurolysis or ablation.
* Coagulation disorders (INR > 1.5, platelet count < 50 × 10⁹/L).
* Severe cardiac, hepatic, or renal insufficiency (Child-Pugh Class C, estimated glomerular filtration rate (eGFR) < 30 mL/min, NYHA Class III-IV heart failure).
* Contraindications to celiac plexus block (e.g., local infection, anatomical variation).
* Any other condition that, in the investigator's judgment, would preclude safe participation in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will enroll adult patients with histologically confirmed advanced biliary tract cancer or pancreatic cancer, who are experiencing moderate to severe cancer-related abdominal pain and are candidates for first-line systemic therapy combined with celiac plexus neurolysis for pain management. Key inclusion criteria involve specific pain intensity, performance status, and organ function requirements.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Estimated)
Dates: Start 2025-12-26 (Actual); Primary Completion 2028-06-26 (Estimated); Study Completion 2028-12-26 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From the start of combination therapy until the first documented disease progression or the end of follow-up, assessed up to 2 years.
  The proportion of participants achieving a best overall response of Complete Response (CR) or Partial Response (PR) according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) during the period from the start of first-line systemic therapy combined with celiac plexus neurolysis (CPN) until disease progression or the end of follow-up (up to 2 years). Tumor assessments will be performed via contrast-enhanced CT or MRI scans at baseline and every 8-12 weeks thereafter.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From the start of combination therapy until the first documented progression or death from any cause, assessed up to 2 years.
  The time from the start of combination therapy to the first documented disease progression according to RECIST 1.1 or death from any cause, whichever occurs first. The median PFS and its 95% confidence interval (CI) will be estimated using the Kaplan-Meier method. PFS rates at 6, 9, and 12 months will be calculated and compared using the stratified log-rank test. Hazard ratios and 95% CIs will be estimated using a stratified Cox proportional hazards model.
Overall Survival (OS) | From the start of combination therapy until death from any cause, assessed up to 3 years.
  The time from the start of combination therapy to death from any cause.
Change in Pain Intensity (Numerical Rating Scale, NRS) | Baseline, and at 4, 8, and 12 weeks after the start of combination therapy.
  The change in the 11-point Numerical Rating Scale (NRS) score for average abdominal pain intensity (ranging from 0 [no pain] to 10 [worst pain imaginable]) from baseline to 4, 8, and 12 weeks after the initiation of combination therapy. A negative change indicates pain reduction. Comparisons will be made using paired t-tests.
Change in Quality of Life (QoL) Scores (EORTC QLQ-C30) | Baseline, and at 12 and 24 weeks after the start of combination therapy.
  The change in the global health status / quality of life scale scores of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) from baseline to 12 and 24 weeks after the initiation of combination therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No